CLINICAL TRIAL: NCT06972732
Title: A Randomized, Open-label, Active-controlled, Parallel, Multicenter, Phase IV Clinical Trial to Compare the Efficacy and Safety of Switching Metformin+SGLT2-i+Dipeptidyl Peptidase-4-inhibitor(DPP-4-i) to Metformin+SGLT2-i+TZD in Patients With Type 2 Diabetes
Brief Title: A Phase IV Clinical Trial to Compare the Efficacy and Safety of Metformin+Sodium-Glucose Cotransporter 2 Inhibitor(SGLT2-i)+Thiazolidinedione (TZD) in Patients With Type 2 Diabetes
Acronym: TELOS
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Boryung Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BR-DPC-CT-401
Record Dates: First submitted 2025-05-07; First posted 2025-05-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Type 2 Diabetes
Keywords: type 2 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Metformin; dapagliflozin; Pioglitazone; Sitagliptin Phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Metformin + Dapagliflozin 10mg/Pioglitazone 30mg (Experimental): One tablet of Metformin and one tablet of Dapagliflozin 10mg/Pioglitazone 30mg administered orally once daily for 24 weeks.
  Interventions: Drug: Metformin; Drug: Dapagliflozin/Pioglitazone
- Metformin + Dapagliflozin 10mg/Sitagliptin 100mg (Active Comparator): One tablet of Metformin and one tablet of Dapagliflozin 10mg/Sitagliptin 100mg administered orally once daily for 24 weeks.
  Interventions: Drug: Metformin; Drug: Dapagliflozin/Sitagliptin

INTERVENTIONS:
Drug: Metformin — The dosage and dose frequency are maintained as they were before the screening.
Drug: Dapagliflozin/Pioglitazone — Dapagliflozin 10mg/Pioglitazone 30mg QD
  Arms: Metformin + Dapagliflozin 10mg/Pioglitazone 30mg
Drug: Dapagliflozin/Sitagliptin — Dapagliflozin 10mg/Sitagliptin 100mg QD
  Arms: Metformin + Dapagliflozin 10mg/Sitagliptin 100mg

SUMMARY:
This is a randomized, open-label, active-controlled, parallel, multicenter, phase IV clinical study evaluating the efficacy and safety of switching Metformin+SGLT2-i+DPP4-i to Metformin+SGLT2-i+TZD in patients with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Has voluntarily agreed to participate in this clinical trial.
* Adults over 19 years of age
* Diagnosed with type 2 diabetes

Exclusion Criteria:

* Has severe renal and liver disorders
* Has type 1 diabetes
* Those who are participating or have participated in other clinical trials and administered their investigational products within 8 weeks before the screening date for this study
* Those who are deemed ineligible to participate in the study by the investigator

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Estimated)
Dates: Start 2025-06-11 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
HbA1c (%) change at 24 weeks compared to the baseline (Visit 2) | From baseline to end of treatment at 24 weeks
  The mean change of HbA1c at 24 weeks compared to the baseline (Visit 2) is evaluated.

CONTACTS AND LOCATIONS:
Locations (1):
- The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul, Seocho District, South Korea

IPD SHARING:
Plan to Share IPD: No